CLINICAL TRIAL: NCT01806831
Title: Efficacy and Safety of Biocellulose Sheet From Coconut Juice Containing Anti-hyperpigmentation Agent ("Biocellulose Mask", "Farhorm®") in Patients Receiving Laser Treatment
Brief Title: Efficacy and Safety of Biocellulose Sheet Containing Anti-hyperpigmentation Agent ("Biocellulose Mask", "Farhorm®") in Patients Receiving Laser Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: Agricultural Research Development Agency (Public Organization) (Unknown)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Associate Professor, Chulalongkorn University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CU 12-33-009
Record Dates: First submitted 2013-03-05; First posted 2013-03-07 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Skin Pigmentation; Skin Irritation
MeSH Terms: conditions — Pigmentation Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: "Biocellulose Mask", Farhorm®"

SUMMARY:
The laser areas treated with biocellulose sheet from coconut juice containing anti-hyperpigmentation agent ("biocellulose mask", "Farhorm®") heal faster than vaseline ointment which is a standard treatment.

DETAILED DESCRIPTION:
Volar surface at upper arm (2X2 cm) on both sides were treated with semi ablative, 1,550 nm Erbium: glass fractional laser. Biocellulose sheet from coconut juice containing anti-hyperpigmentation agent ("biocellulose mask","Farhorm®")was applied for 20 min on one side and the other side was treated with vaseline ointment. The redness, skin hydration and skin pigmentation were evaluated at that area before laser, immediately after laser and after applying the treatment. These parameters were compared between treatment (area treated with Biocellulose sheet from coconut juice containing anti-hyperpigmentation agent, "biocellulose mask", "Farhorm®") and control (vaseline ointment).

ELIGIBILITY:
Inclusion Criteria:

* Age 20-50 years old
* No skin problem such as inflammation, fresh wounds
* Not receive laser treatment during last 3 months
* No history of smoking or alcohol drinking
* No allergy to licorice extract, Vit C, Vit E, arbutin or stearyl glycyrrhetinate
* Willing to participate in this study and can comply with study protocol

Exclusion Criteria:

* Has history of hyperallergic reaction
* Has wound(s) on face during last 4 weeks
* Has history of eczema, psoriasis during last 6 months
* Has laser treatment during last month
* Use steroid, antibiotic, anti-inflammatory drugs or antihistamine during 3 days before recruiting
* Had major surgery during last 12 months
* Has history of cancer during last 12 months
* Pregnant or lactation

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-09; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The skin pigmentation immediately after laser therapy and after using biocellulose mask | Change from immediately after laser treatment and 30 min after laser and treatment with mask

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pharmacy Practice, Faculty of Pharmaceutical Sciences, Chulalongkorn Unviersity, Bangkok, Bangkok, Thailand